CLINICAL TRIAL: NCT02830776
Title: Topical Bimatoprost for Chemical Blepharoplasty
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 833277-1
Record Dates: First submitted 2016-07-07; First posted 2016-07-13 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Dermatochalasis
Keywords: dermatochalasis; bimatoprost; blepharoplasty
MeSH Terms: conditions — Cutis Laxa | interventions — Bimatoprost; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): This is a single-arm open label proof of concept pilot study evaluating use of Latisse (bimatoprost 0.03% ophthalmic solution) applied to the eyelid margin for dermatochalasis (upper eyelid drooping).
  Interventions: Drug: bimatoprost 0.03% ophthalmic solution

INTERVENTIONS:
Drug: bimatoprost 0.03% ophthalmic solution — Latisse (bimatoprost 0.03% ophthalmic solution) applied to the eyelid margin for dermatochalasis (upper eyelid drooping)
  Other Names: Latisse

SUMMARY:
Topical bimatoprost has been shown to cause periorbital changes of soft tissue which are most pronounced when used directly onto the cornea for the treatment of glaucoma. Changes are primarily felt to be the result of prostaglandin-mediated adipocyte loss, resulting in deepening of the upper eyelid sulcus and recession of infraorbital pseudoherniation. Use of topical bimatoprost to the upper eyelid margin, now FDA approved for eyelash enhancement, may provide a metered effect on the periocular tissues and allow for a topical approach to periocular rejuvenation.

This is a proof of concept study which aims to enroll a series of patients with mild to severe dermatochalasis, treat with topical bimatoprost 0.03% solution to the upper lid margin, and evaluate for cosmetic improvement of the periocular area.

DETAILED DESCRIPTION:
Perception of beauty in the periocular region is influenced by several factors, including symmetry, population norms, and skin texture and tone. Soft tissue and skin changes over time create an aged appearance with the development of dermatochalasis, blepharoptosis, lacrimal gland prolapse, and fat prolapse. Techniques for periocular rejuvenation are well established and include soft tissue augmentation, resurfacing, and surgical correction. In May 2015, Sarnoff and Gotkin reported a case of "chemical blepharoplasty" achieved with topical bimatoprost ophthalmic 0.03% solution applied to the upper eyelid margin. After three months of use, the author noted a more youthful appearance of the periocular region, with deepening of the upper eyelid sulcus, reduction in dermatochalasis, and diminution of the inferior eyelid fat pad. These changes were attributed to the prostaglandin associated periorbitopathy (PAP), a well described phenomenon observed with the use of topical prostaglandin analogues use for glaucoma.

Periorbital changes observed with topical prostaglandin analogues are primarily due to effects on aponeurotic and deep orbital adipocytes. Prostaglandins activate the adipocyte mitogen-activated protein kinase (MAPK) pathway, leading to inactivation of peroxisome proliferator-activated receptor (PPAR)-gamma, inhibition of adipocyte differentiation, and decreased fat accumulation within adipocytes. Bimatoprost concentration-dependent contractions of ciliary muscles and activation of matrix metalloproteinases may also contribute to periocular changes. Patients using topical ophthalmic prostaglandin analogues commonly develop periorbital fat loss, which has been well characterized in the ophthalmology literature.

Bimatoprost applied to the upper eyelid margin for eyelash enhancement attempts to capitalize on the desirable effects of darker, longer, thicker eyelashes, while limiting more significant and undesirable effects through limited exposure of the drug to ocular tissues. This same concept may apply for dermatochalasis: at a metered dose, topical bimatoprost to the lid margin could lead to subtle periorbital fat loss resulting in improved dermatochalasis.

ELIGIBILITY:
Inclusion Criteria:

* 18+,
* mild to severe dermatochalasis, desire for enhanced eyelashes.

Exclusion Criteria:

* Patients with current use of ophthalmic prostaglandin analogues,
* history of blepharoplasty,
* history of neuromodulators or fillers to the periocular region or frontalis in the last 6 months,
* existing deep upper eyelid sulcus,
* opposition to eyelash enhancement,
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan P Couvillion, MD, MS, Principal Investigator — Tulane University School of Medicine, Department of Dermatology
Locations (1):
- Tulane Department of Dermatology, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarnoff DS, Gotkin RH. Bimatoprost-induced chemical blepharoplasty. J Drugs Dermatol. 2015 May;14(5):472-7. PMID 25942665
- [Background] Filippopoulos T, Paula JS, Torun N, Hatton MP, Pasquale LR, Grosskreutz CL. Periorbital changes associated with topical bimatoprost. Ophthalmic Plast Reconstr Surg. 2008 Jul-Aug;24(4):302-7. doi: 10.1097/IOP.0b013e31817d81df. PMID 18645437
- [Background] Reginato MJ, Krakow SL, Bailey ST, Lazar MA. Prostaglandins promote and block adipogenesis through opposing effects on peroxisome proliferator-activated receptor gamma. J Biol Chem. 1998 Jan 23;273(4):1855-8. doi: 10.1074/jbc.273.4.1855. PMID 9442016
- [Background] Kucukevcilioglu M, Bayer A, Uysal Y, Altinsoy HI. Prostaglandin associated periorbitopathy in patients using bimatoprost, latanoprost and travoprost. Clin Exp Ophthalmol. 2014 Mar;42(2):126-31. doi: 10.1111/ceo.12163. Epub 2013 Aug 4. PMID 23844550
- [Background] Cohen JL. Enhancing the growth of natural eyelashes: the mechanism of bimatoprost-induced eyelash growth. Dermatol Surg. 2010 Sep;36(9):1361-71. doi: 10.1111/j.1524-4725.2010.01522.x. PMID 20384750
- [Background] Shah M, Lee G, Lefebvre DR, Kronberg B, Loomis S, Brauner SC, Turalba A, Rhee DJ, Freitag SK, Pasquale LR. A cross-sectional survey of the association between bilateral topical prostaglandin analogue use and ocular adnexal features. PLoS One. 2013 May 1;8(5):e61638. doi: 10.1371/journal.pone.0061638. Print 2013. PMID 23650502

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient enrolled in the study but was lost to followup. Data was incomplete for this subject so was not included in final analyses.
Period: Overall Study
Arm/Group | Treatment Group
Started | 15
Completed | 14
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Patients received Latisse (bimatoprost 0.03% ophthalmic solution) applied to the eyelid margin for dermatochalasis (upper eyelid drooping)
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 57 [37 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian | 14
  Ethnicity: African American | 1

OUTCOME MEASURES:

1. Primary Outcome: Graded Change in Dermatochalasis
Description: Patients were followed for 12 weeks total, with visits every 4 weeks for a total of 4 visits. Photodocumentation was performed at each visit. At completion of the study period, each patient's photographs at weeks 0 and 12, were graded by 2 blinded evaluators for level of dermatochalasis: -1 (deep upper eyelid sulcus), 0 (no dermatochalasis), 1 (mild, slightly noticeable), 2 (moderate, noticeable), or 3 (severe, distinctive). The change of dermatochalasis (week 12 score subtracted from week 0 score) was the primary outcome measure. A greater change (based on a higher score) in dermatochalasis indicated better response to the treatment.
Time Frame: At 12 weeks
Population: Patients received Latisse (bimatoprost 0.03% ophthalmic solution) applied to the eyelid margin for dermatochalasis (upper eyelid drooping)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 14
units on a scale | .2679 [0.0970 to 0.4387]

2. Secondary Outcome: Change in Patient Satisfaction
Description: Entry and exit surveys were completed about self perception of the periocular area. The satisfaction was measured based on 2 short surveys. Entry survey had 1 question "how do you rate your satisfaction with your appearance?" - the scale was 0-5, with 0 being "Not at all" to 5 being "extremely." The exit survey posed two questions, (1) "how do you rate satisfaction with your appearance?" with the same 0-5 scale, as well as (2) Do you notice an improvement in your eyelid droop (dermatochalasis)?" with a scale as follows: Worse (-1), No Change (0), 25% better (1), 50% better (2), 75% better (3), or 100% better (4). The change in satisfaction was measured by the summation of scores from both surveys and the average was calculated.
Time Frame: Weeks 0, 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 14
units on a scale | .214 [-.777 to .349]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 7/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=15)
Itching (Skin and subcutaneous tissue disorders) | 5 — Itching at the site of application
Eyelid skin redness (Skin and subcutaneous tissue disorders) | 4
Eyelid darkening (Skin and subcutaneous tissue disorders) | 3
Unexpected hair growth (Skin and subcutaneous tissue disorders) | 1 — Facial pigmented hair growth beyond the eyelashes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT02830776/Prot_000.pdf
  • Informed Consent Form (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/76/NCT02830776/ICF_001.pdf